CLINICAL TRIAL: NCT00074529
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of MK-0677 25 mg in Slowing the Progression of Alzheimer's Disease
Brief Title: Study of MK0677 for the Treatment of Alzheimer's Disease (0677-030)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 0677-030; Formally-BG0812AZ; MK0677-030; 2006_412
Record Dates: First submitted 2003-12-15; First posted 2003-12-16 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ibutamoren mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0677

SUMMARY:
An investigational drug (MK0677) will be studied to determine whether it helps the memory and cognition of patients with Alzheimer's Disease.

ELIGIBILITY:
* Patients must have probable Alzheimer's disease of mild or moderate severity.
* A brain scan and laboratory results must be consistent with Alzheimer's disease.
* The patient must be otherwise medically healthy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2003-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Cognitive function over 12 month period; safety and tolerability | over 12 month period

SECONDARY OUTCOMES:
AD symptoms over a 6 month and 12 month period measured by the CIBIC + and the ADAS-Cog. | over a 6 month and 12 month period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Sevigny JJ, Ryan JM, van Dyck CH, Peng Y, Lines CR, Nessly ML; MK-677 Protocol 30 Study Group. Growth hormone secretagogue MK-677: no clinical effect on AD progression in a randomized trial. Neurology. 2008 Nov 18;71(21):1702-8. doi: 10.1212/01.wnl.0000335163.88054.e7. PMID 19015485
- [Derived] Sevigny JJ, Peng Y, Liu L, Lines CR. Item analysis of ADAS-Cog: effect of baseline cognitive impairment in a clinical AD trial. Am J Alzheimers Dis Other Demen. 2010 Mar;25(2):119-24. doi: 10.1177/1533317509350298. PMID 19949163